CLINICAL TRIAL: NCT06247878
Title: Sleep Apnea Detection and Sleep Staging Using Skiin Wearable Textile Sensors
Brief Title: Skiin-PSG Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Myant Medical Corp. (Industry)
Collaborators: Jodha Tishon Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: PSG-Myant 157487
Record Dates: First submitted 2024-01-09; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: wearable electronic devices; digital health; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep apnea/hypopnea detection: Ability of Skiin underwear chest band in detecting sleep apnea or hypopnea will be tested against polysomnography.
  Interventions: Device: Skiin underwear chest band

INTERVENTIONS:
Device: Skiin underwear chest band — Participants will be asked to wear a skiin underwear chest band during a polysomnography test.

SUMMARY:
The goal of this observational study is to develop new algorithms to detect apnea and/or hypopnea to provide additional insights to Skiin users and to their circle of care to validate and/or improve the current algorithms of the Skiin system for extraction of biological metrics during sleep based on the Skiin ECG and accelerometry data.

DETAILED DESCRIPTION:
Eligible individuals who consent to participate will be asked to wear a Skiin Underwear chest band while going through a polyssomnography test.

1. Investigational device

   The Skiin underwear chest band is worn at the under-chest level (under the pectoral or breast fold), and is connected to the Skiin Connected Life App (SCLA). The app collects ECG, accelerations, and temperature to generate metrics such as sleep, activity, and other physiological biometrics (resting heart rate, heart rate variability, breathing rate). The investigator will ensure the chest band is worn properly as defined by the vertical line on the band besides the Skiin logo corresponding with the center of the body.
2. Polysomnography

The equipment being used for polysomnography is the Embla Sandman Elite PSG System. In advance to the test, patients receive information about the PSG test procedure and patients are usually instructed to avoid naps and stimulants (i.e., caffeine) during the day of the test. A list of instructions is usually provided to the patient.

Once the patient is ready for bed, the technologists will place sensors on the patient's scalp, temples, chest and legs using a mild adhesive, such as glue or tape. The sensors are connected by wires to a computer (wires are long enough to let the patient move around in bed). A small clip is placed on the finger or ear to monitor the level of oxygen in the blood.

Electrodes location - monitoring location includes:

* Electroencephalography (EEG) - The placement of the EEG electrodes on the scalp follows an international system known as the 10-20 system of electrode placement. This is a standardized method of identifying equally spaced electrode positions on the scalp, based on four identifiable skull landmarks.
* Electromyography (EMG) - Chin EMG records muscle tone at the mentalis and submentalis muscles. For the leg EMG two electrodes are placed about 2 to 4 cm apart longitudinally, along the belly of the anterior tibialis muscle of each leg, to record periodic limb movements.
* Electrooculography (EOG) - to record rapid eye movements of REM sleep and to assess sleep onset.
* Electrocardiography (ECG) - gel electrodes applied to the right and left subclavicular areas (essentially lead I) or the right subclavicular area and the lower left thorax (essentially lead II).
* Airflow (nasal/oral) - thermal sensors or pressure sensing
* Pulse oximetry - oximeter placed on the index finger
* Respiratory effort (thoracic/abdominal) - belts placed around the chest and abdomen to monitor movements.
* Snore sensor - small microphone
* Body position - monitoring with sensors

Bio-calibration - is a series of actions that the patient is asked to perform before initiating the PSG test. This is to ensure that the sensors are measuring what they are supposed to and to verify signal quality.

Audio-visual recording - video and audio recording is part of the clinic's standard PSG test. It allows the clinician to observe the patient's behavior during the sleep study to improve clinical interpretation and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred to do a polysomnography
* Diagnosed or suspected obstructive sleep apnea (OSA)
* 18 years old or more
* Understand and speak English enough to consent

Exclusion Criteria:

* Pregnant women
* Implanted defibrillator or pacemaker
* Absence of a garment fitting the participant's body
* An open wound or dressing (e.g. band-aid) on a body part that needs to be in contact with the Skiin electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit 200 individuals > 18 years old, referred to a polysomnography test due to a diagnosed or suspected obstructive sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Skiin system for detection of apnea/hypopnea compared to Polysomnography | Over one night, 8 to 12 hours total
  Apnea/hypopnea events identified in the Skiin system will be compared to Apnea/hypopnea events identified in the polysomnography system. Data will be categorized as true positive, false positive, false negative to calculate the sensitivity, specificity, PPV, NPV).

SECONDARY OUTCOMES:
Accuracy of Skiin system for detection of sleep duration compared to Polysomnography | Over one night, 8 to 12 hours total
  Sleep duration recorded by the Skiin system will be compared to Sleep duration recorded by the Polysomnography system to assess accuracy. Differences, bias, and Root Mean Square Error will be calculated for each participant and for the group.
Accuracy of Skiin system for estimation of breathing rate compared to Polysomnography | Over one night, 8 to 12 hours total
  Resting breathing rate calculated by the Skiin system over night will be compared to resting breathing rate calculated by the Polysomnography for accuracy check.
  Differences, bias, and Root Mean Square Error will be calculated for each participant and for the group.
Accuracy of Skiin system for calculation of resting heart rate compared to Polysomnography | Over one night, 8 to 12 hours total
  Resting heart rate calculated by the Skiin system over night will be compared to resting heart rate calculated by the polysomnography for accuracy check.
  Differences, bias, and Root Mean Square Error will be calculated for each participant and for the group.
Accuracy of Skiin system for calculation of heart rate variability compared to polysomnography | Over one night, 8 to 12 hours total
  Heart rate variability (RMSSD) calculated by the Skiin system over night will be compared to heart rate variability calculated based on the polysomnography system's data.
  Differences, bias, and Root Mean Square Error will be calculated for each participant and for the group.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Shapiro, MD, Principal Investigator — Jodha Tishon
Locations (1):
- International Sleep Clinic WPSHC, Parry Sound, Ontario, Canada